CLINICAL TRIAL: NCT01748422
Title: The Role of Qutenza (Topical Capsaicin 8%) in Treating Neuropathic Pain From Arteriovenous Fistulae in Patients With End Stage Renal Failure
Brief Title: Qutenza (Topical Capsaicin 8%) for Painful Arteriovenous Fistulae
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Dr Patrick Kearns, Principal Investigator, NHS Greater Glasgow and Clyde
Other Study IDs: GU11SB126
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Neuropathic Pain; Arteriovenous Fistulae
Keywords: Neuropathic pain; Arteriovenous fistulae; End stage renal disease
MeSH Terms: conditions — Neuralgia; Kidney Failure, Chronic | interventions — Capsaicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental: Qutenza: Single treatment with Qutenza (topical capsaicin8%) transdermal patch
  Interventions: Drug: Qutenza

INTERVENTIONS:
Drug: Qutenza — Transdermal patch
  Other Names: Topical capsaicin 8%

SUMMARY:
Arteriovenous fistulae are artificial connections between the artery and vein in the arm which allow needles to be inserted for haemodialysising patients wit kidney failure. Occasionally severe debilitating pain can arise from these fistulae for which no cause can be found. Such pain can be very difficult to treat. Many commonly used used painkillers are known to cause significant side effects in patients with renal failure (drowsiness, confusion etc.

Qutenza (topical capsaicin 8%) is a new treatment made from chilli peppers which is applied to the skin as a patch and works directly at the nerve endings in the skin to prevent pain. It therefore should not have the systemic side effects of other drugs. It has been demonstrated to be beneficial in other painful conditions for example post-shingles pain and nerve pain from HIV. It has never been used for critical ischaemia before.

We propose to investigate the efficacy of Qutenza in treating patients with end stage renal failure and chronic pain from their fistulae (AVF). We will recruit 20 patients with painful AVF and treat them with Qutenza. We will follow them up for 12 weeks and monitor the change in their pain scores.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients >18 years old with end stage renal disease on dialysis and significant chronic neuropathic pain arising from their arteriovenous fistula (defined as pain with symptoms to suggest a neuropathic element occurring most days for at least a month which has not responded to simple analgesia)

Exclusion Criteria:

* Pre-dialysis
* Underlying anatomical/ structural abnormality with AVF contributing to pain
* Diabetic neuropathy resulting in sensory loss
* Hypersensitivity to Qutenza, Emla or any of the excipients
* Broken skin or active ulceration at the site of application
* Severe uncontrolled hypertension (systolic BP >200)
* Proven cardiac event during the preceding 3 months
* Women who are pregnant or breast feeding
* Lack of capacity or inability to provide informed consent
* Declines participation in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage renal failure and chronic neuroapthic pain arising fromt heir arteriovenous fistulae
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain | 12weeks
  As assessed by Visual Analogue Pain Score

SECONDARY OUTCOMES:
Neuropathic pain | 1 week, 6 weeks
  As assessed by Visual Analogue Pain Score and Brief Pain Inventory
Quality of life | 6 weeks, 12 weeks
  As assessed by EQ-5D
Safety and tolerability | 1 week, 6 weeks and 12 weeks
  As assessed by: Number of adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick K Kearns, MBChB, Principal Investigator — NHS Greater Glasgow and Clyde; Marc Clancy, FRCS, PhD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Department of Renal Surgery, Queen Elizabeth University Hospital, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided